## **Encouraging Healthy and Sustainable Dietary Substitutions**

NCT06175026

September 22, 2023

## STANFORD UNIVERSITY Research Information Sheet

Protocol Director: Anna Grummon

Protocol Title: Dietary messages

IRB Use Only

Approval Date: September 22, 2023

Expiration Date: Does not expire

**DESCRIPTION:** You are invited to participate in a research study on your reactions to different messages. The purpose of the research is to understand how adults react to different messages. In this survey, you will be asked to view a variety of messages and respond to questions asking about your reaction to those messages. We are asking for your permission to tell you exactly what we are studying once the research has ended. Participation in this research is voluntary, and you are free to withdraw your consent at any time.

The National Institutes of Health are providing financial support for this study.

**TIME INVOLVEMENT:** Your participation will take approximately 8-10 minutes.

**RISKS AND BENEFITS:** The risks associated with this study are accidental disclosure of the data collected during the survey, however this is very unlikely given the steps in place to reduce this risk. We will take several steps to reduce the risk of accidental disclosure. First, we will not collect any health information or individually identifiable information. Second, we will store all study data in a password-protected server. Third, only the study team will have access to the raw data. Fourth, all staff will be trained in proper handling of participant data. We cannot and do not guarantee or promise that you will receive any benefits from this study.

**PAYMENTS:** You will receive the amount and type of payment for your participation as displayed in the invitation you received to participate in this study.

**PARTICIPANT'S RIGHTS:** If you have read this form and have decided to participate in this project, please understand your participation is voluntary and you have the right to withdraw your consent or discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled. The alternative is not to participate. You have the right to refuse to answer particular questions. The results of this research study may be presented at scientific or professional meetings or published in scientific journals. Your individual privacy will be maintained in all published and written data resulting from the study. Identifiers might be removed from identifiable private information and, after such removal, the information could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you.

## **CONTACT INFORMATION:**

Questions: If you have any questions, concerns, or complaints about this research, its procedures, risks and benefits, contact the Protocol Director, Dr. Anna Grummon at (650)644-7366 or agrummon@stanford.edu.

Independent Contact: If you are not satisfied with how this study is being conducted, or if you have any concerns, complaints, or general questions about the research or your rights as a participant, please contact the Stanford Institutional Review Board (IRB) to speak to someone independent of the research team at 650-723-5244 or toll free at 1-866-680-2906. You can also write to the Stanford IRB, Stanford University, 1705 El Camino Real, Palo Alto, CA 94306.

Please print a copy of this page for your records.

If you agree to participate in this research, please click "I consent."